CLINICAL TRIAL: NCT06918873
Title: Quality of Life During Different Regimens of Combined Hormonal Contraceptives in Women of Reproductive Age
Status: Recruiting | Type: Observational
Sponsor: Fondazione IRCCS Policlinico San Matteo di Pavia (Other)
Responsible Party: Principal Investigator, Rossella Nappi, Principal Investigator, Fondazione IRCCS Policlinico San Matteo di Pavia
Other Study IDs: REN13
Record Dates: First submitted 2025-03-26; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Hormonal Contraception
Keywords: combined hormonal contraception; female sexual dysfunction; mood disorders
MeSH Terms: conditions — Mood Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The aim of the present study is to investigate the psychosexual effects of combined hormonal contraception regimens, comparing them in terms of estrogen type and dosage, hormonal combination regimen and different routes of administration, in women seeking a hormonal contraception method to prevent unwanted pregnancies. In particular, the study focuses on the incidence of mood disorders and sexual dysfunctions associated with distress in the entire study population using combined hormonal contraception. It will also examine the incidence of these conditions under the influence of specific combined hormonal contraceptives, as well as whether different types of progestins and the route of administration (oral, vaginal or transdermal) may affect the occurrence of mood disorders and sexual dysfunctions.

ELIGIBILITY:
Inclusion Criteria:

* women of childbearing age (aged 18-40) who seek advice for use of combined hormonal contraception (CHC).
* stable relationship

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Study Population: Women referred for prescription of a hormonal contraceptive.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2014-05-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Impact of different estrogen-progestin contraception regimens on sexual function and sexually related distress. | 6 months
  Evaluate the trend of the scores of the Female Sexual Function Index (FSFI) in the entire study population using combined hormonal contraception (CHC), both at baseline and after 6 months of CHC exposure; evaluate whether the FSFI scores vary significantly in relation to the type and dosage of estrogen used in hormonal contraception; evaluate the extent of female sexual distress score (FSDS) in the entire study population using CHC, both at baseline and after 6 months of CHC exposure; evaluate whether the FSDS scores vary significantly in relation to the type and dosage of estrogen used in hormonal contraception.

SECONDARY OUTCOMES:
Impact of combined hormonal contraception on mood disorders | 6 months
  Evaluate mood disorders (Hospital Anxiety and Depression score [HADS] > 10) in the entire study population taking CHC, at baseline and after 6 months of CHC exposure; evaluate if there are significant differences in the onset mood disorders based on the type of estrogen, its dosage, the pharmacological class of the progestin, and the type of contraceptive administration (oral, vaginal, transdermal).
Impact of basal clinical variables mood disorders and sexual dysfunction in women using combined hormonal contraception | 6 months
  Evaluate if certain basal characteristics of menstrual cycles, psychological well-being and quality of life (assessed through validated questionnaires) are correlated with the extent of sexual dysfunctions (FSFI, FSDS) and mood (HADS) both at baseline and after 6 months of CHC therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione IRCCS Policlinico San Matteo, SSD Ostetricia e Ginecologia 2 - Riproduzione e Procreazione Medicalmente Assistita, Pavia, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No